CLINICAL TRIAL: NCT01276717
Title: Phase I Trial of Carfilzomib (PR-171) in Combination With Vorinostat (SAHA) in Patients With Relapsed/Refractory B-Cell Lymphomas
Brief Title: Study of Carfilzomib and Vorinostat for Relapsed or Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Massey Cancer Center (Other)
Responsible Party: Principal Investigator, Jonathan Friedberg, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32833
Record Dates: First submitted 2010-11-10; First posted 2011-01-13 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — carfilzomib; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat + Carfilzomib (Experimental)
  Interventions: Drug: Drug: Carfilzomib; Drug: Vorinostat

INTERVENTIONS:
Drug: Drug: Carfilzomib — Carfilzomib 30 minutes infusion daily for days 1, 2, 8, 9, 15, 16, Every 28 days. A maximum of 13 cycles will be administered.
  Other Names: PR-171
Drug: Vorinostat — Vorinostat by mouth twice daily on days 1, 2, 3, 8, 9, 10, 15, 16 and 17. Maximum 13 cycles.
  Other Names: Zolinza®

SUMMARY:
This will be a phase I study of carfilzomib in combination with vorinostat in patients with relapsed/refractory B-cell lymphomas. Combination therapy with proteosome inhibitor PR-171 and HDAC inhibitors is highly synergistic in primary DLBCL cells, and both classes of drugs can also synergize powerfully to induce cell death in bortezomib-resistant cells. The purpose of this study is to see if vorinostat can combine with carfilzomib and to safely find the recommended phase II dose.

DETAILED DESCRIPTION:
Study Drugs:

Vorinostat, a class I/II pan-histone deacetylase inhibitor (HDACI), was the first approved agent og this class on the basis of activity in refractory cutaneous T-cell Lymphoma. Lethal mechanisms include anti-apoptotic protein down-regulation, up-regulation of proapoptotic proteins, induction of ROS, death receptor up-regulation, and disruption of chaperone function and DNA-repair proteins.

Carfilzomib, is a irreversible proteasome inhibitor of the epoxyketone class that exhibits a high level of selectivity for the proteosome. This agent induced a dose- and time-dependent inhibition of proliferation, ultimately leading to apoptosis.

Study Drug Administration:

If you are found to be eligible to take part in this study:

* Vorinostat PO twice daily on Days 1, 2, 3, 8, 9, 10, 15, 16 and 17.
* Daily Carfilzomib 30 minutes infusion on Days 1, 2, 8, 9, 15, 16.
* Administer first daily dose of vorinostat prior to carfilzomib on Days 1, 2, 8, 9, 15, 16
* Cycle repeated every 28 days, up to 13 cycles.

Carfilzomib will be given at 20mg/m2 for days 1 and 2 of cycle 1 only, then escalated to the higher dose indicated in the schema on day 8 of cycle 1 and thereafter. Carfilzomib treatment is to be done early in the morning and have a minimum of a 6 hour observation period after the infusion. For patients with good tolerability to carfilzomib during the first cycle, an observation period of 2 hours is recommended. A minimum of 16 hours should separate doses of carfilzomib, so that the day 1 dose may be given in the afternoon and the day 2 dose in morning during cycle 2 and subsequent cycles for patients who tolerate the drug well.

If two out of 6 patients do not tolerate the initial dose of 20 mg/m2 carfilzomib on days 1 & 2 followed by 27 mg/m2 carfilzomib for subsequent doses and 200 mg/day bid vorinostat, the next patient should be dose reduced to 20 mg/m2 carfilzomib and 100 mg/day bid vorinostat.

Study Visits:

* Baseline within 4 weeks of Cycle 1 Day 1.
* CT or physical exam.
* Bone marrow if needed to follow disease status.
* PET recommended but not required. To document complete response (CR), a PET is REQUIRED.
* Optional research tumor biopsy.
* Peripheral blood obtained for PD prior to initiation of treatment and at 48 hours +/- 6 hours after receiving first dose of Carfilzomib , and at Off Study.
* End of Treatment Restaging will take place 6-8 weeks after completion of treatment and will include an assessment by the physician, labs, and a tumor response evaluation.
* After completion of Restaging exams, Follow up exams will take place every 6 months for 2 years and then annually until disease progression or initiation of another treatment.
* An Off Study visit will take place at the time of disease progression or initiation of another treatment, which will include assessment by the physician,a tumor response evaluation, labs, and a final PD sample, by the patient's consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell lymphomas, excluding CLL (Chronic Lymphocytic Leukemia), that is recurrent or refractory after at least one prior therapy and for which no other potentially curative therapy is available.
* Age ≥ 18 years
* ECOG Performance Status (PS) ≤ 2
* Laboratory parameters

  * if SLL, lymphocyte count < 5,000/µL
  * Absolute neutrophil count ≥ 1000/µL
  * Platelets ≥ 75,000/µL
  * Creatinine ≤ 1.5x upper limit of normal or calculated creatinine clearance > 40mL/min
  * AST, ALT ≤ 2.5 x upper limit of normal (ULN)
  * Bilirubin ≤ 2.0 mg/mL
  * Serum potassium ≥ 3.5 mEq/L and serum magnesium ≥ 1.7 mEq/dL (electrolytes may be corrected with supplementation).
  * PT < 1.5 x ULN and PTT < 1.2 x ULN (unless receiving therapeutic anticoagulation).
* Patient is, in investigator's opinion, willing and able to comply with the protocol requirements and offers written informed consent.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control ( i.e., oral injectable hormonal methods; barrier methods such as intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence)for the duration of the study.
* Male subject agrees to use an acceptable method for contraception for the duration of study.

Exclusion Criteria:

* History of brain metastasis including leptomeningeal metastasis.
* Chemotherapy of radiotherapy within 3 weeks prior to entering the study.
* Prior histone deacetylase inhibitor as cancer treatment.
* Concurrent treatment with other investigational agents or cancer treatment.
* Unable to take oral medications.
* Active ischemic heart disease or congestive heart failure. If there is suspicion of cardiac disease, left ventricular ejection fraction (LVEF) must be ≥ 45%, otherwise study to evaluate EF is not required.
* Persistent blood pressure (BP) of ≥ 160/95 (three separate readings on different days).
* History of allergic reactions attributed to compounds of similar chemical or biological composition to carfilzomib and vorinostat.
* Known clinical significant infection including infection with human immunodeficiency virus (HIV), or active hepatitis B or C, requiring treatment.
* Serious medical or psychiatric illness likely to interfere with patient participation.
* Pregnant or nursing. Confirmation that a woman is not pregnant must be established by a negative serum pregnancy test result obtained at screening.
* Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* No prior allogeneic stem cell transplant.
* Patients scheduled for any type of stem cell transplant within 4 weeks of treatment.
* Patients who have valproic acid for epilepsy can enroll, provided that they stopped drug at least 30 days prior to enrollment and they will be on a stable, effective dose of an alternative anti-seizure medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants who experience Adverse Events as a Measure of Safety and Tolerability | From date of study entry until the 30 days after the last dose of study treatment.
  Determine the recommended phase II doses for the combination of carfilzomib and vorinostat in patients with relapsed or refractory B cell lymphoma.

SECONDARY OUTCOMES:
Number of Participants who Respond to Treatment | From the date of completion of first cycle of treatment until the date of best response to treatment, as determined by restaging scans
  Determine response rate to combination of carfilzomib and vorinostat.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Friedberg, M.D., Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - University of Rochester, Rochester, New York
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia